CLINICAL TRIAL: NCT03636529
Title: Anthocyanin-rich Tart Cherry Juice Consumption and Reduced Biomarkers of Inflammation, CVD, and Diabetes.
Brief Title: Tart Cherry Juice and Markers of Inflammation, CVD, and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Keith Martin, Research Assistant Professor, University of Memphis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 0902003690
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Hyperuricemia; Insulin Resistance; Obesity; CVD
Keywords: obese; overweight; tart cherry juice
MeSH Terms: conditions — Hyperuricemia; Insulin Resistance; Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: In this study, the investigators recruited at-risk individuals who were overweight (25.0-29.9 kg/m2) and obese (> 30.0 kg/m2) and likely to exhibit one or more conditions associated with MetS. In this 12-week placebo-controlled 2 x 2 crossover dietary intervention, the investigators randomized participants to consume 240 mL (8 ounces) daily of either placebo (artificial cherry-flavored, anthocyanin-free beverage) or TCJ for 4 weeks, followed by a 4-week washout period, then consumption of the alternate beverage for 4 weeks. Subsequently, the investigators determined the effect of TCJ in at-risk participants on markers of uricemia, lipidemia, glycemia, and inflammation.
Who Masked: Participant
Masking Description: Placebo beverage was prepared in the ASU metabolic kitchen and matched for fructose and total carbohydrate concentrations as well as being artificially colored to match tart cherry juice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tart cherry juice (TCJ) (Active Comparator): Participants randomized to consume either placebo beverage or tart cherry juice at beginning of the study followed by a 4 week washout then switch over to the alternate beverage to account for timing and order effects.
  Interventions: Dietary Supplement: Tart cherry juice
- Placebo (Placebo Comparator): Participants randomized to consume either placebo beverage or tart cherry juice at beginning of the study followed by a 4 week washout then switch over to the alternate beverage to account for timing and order effects.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Tart cherry juice — Participants randomized to consume for 4-weeks either placebo beverage or single-strength tart cherry juice at beginning of the study followed by a 4 week washout then switch over to the alternate beverage for 4 weeks to account for timing and order effects.
  Arms: Tart cherry juice (TCJ)
Other: Placebo — Participants randomized to consume either placebo beverage or tart cherry juice at beginning of the study followed by a 4 week washout then switch over to the alternate beverage to account for timing and order effects.
  Arms: Placebo

SUMMARY:
In this study, the investigators recruited at-risk individuals (n=26) who were overweight (25.0-29.9 kg/m2) and obese (> 30.0 kg/m2) and likely to exhibit one or more conditions associated with Metabolic Syndrome (MetS). In this 12-week placebo-controlled 2 x 2 crossover dietary intervention, the investigators randomized participants to consume 240 mL (8 ounces) daily of either placebo (artificial cherry-flavored, anthocyanin-free beverage) or TCJ for 4 weeks, followed by a 4-week washout period, then consumption of the alternate beverage for 4 weeks. Subsequently, the investigators determined the effect of TCJ in at-risk participants on markers of uricemia, lipidemia, glycemia, and inflammation.

DETAILED DESCRIPTION:
In this study, the investigators recruited at-risk individuals (n=26) who were overweight (25.0-29.9 kg/m2) and obese (> 30.0 kg/m2) and likely to exhibit one or more conditions associated with MetS. Participants were >18 years of age, not pregnant, not diabetic, with no unresolved infections or diseases (diabetes, CVD, IBD, cancer and liver disease), and nonsmokers. Histories of medication and dietary supplement use were collected and those taking anti-inflammatory or lipid-lowering medications were excluded. After enrollment, participants were randomly assigned to consume daily either 240 mL (8 ounces) of TCJ diluted (1:6 v/v) from concentrate (Coloma Frozen Foods, Coloma, MI ) or a placebo beverage for 4 weeks. The placebo was prepared by combining 48.3 g each of dextrose and fructose (Batory Foods, Des Plaines, IL), food-grade red and blue dyes (2.0 mL and 0.1 mL, respectively; McCormick & Company, Inc., Sparks, MD), lemon powder drink mix (0.8 g; True Citrus, Baltimore, MD), powdered black cherry drink mix (4.0 g; Kraft Foods Group, Inc., Northfield, IL), and filtered, bottled water (local supermarket) to produce 1 liter of placebo beverage. After a 4-week washout period, participants consumed the alternate beverage for 4 weeks in this 12-week 2x2 crossover, placebo-controlled dietary intervention. Subsequently, the investigators determined the effect of TCJ in at-risk participants on markers of uricemia (sUA), lipidemia (HDL, LDL, triglycerides, VLDL, total cholesterol), glycemia (fasting insulin and glucose, HOMA, QUICKI, McAuley indirect indices), and inflammation (hsCRP, TNF-alpha, and ESR).

ELIGIBILITY:
Inclusion Criteria:

* This study was a 12-week 2 x 2 crossover, randomized, placebo-controlled dietary intervention in overweight and obese participants (BMI>25.0 kg/m2) who are more likely to exhibit >1 of the 5 risk conditions associated with metabolic syndrome (MetS). BMI was the minimal criterion for recruitment.

Exclusion Criteria:

* Participants were >18 years of age, not pregnant, not diabetic, with no unresolved infections or diseases (diabetes, CVD, IBD, cancer and liver disease), and nonsmokers. Histories of medication and dietary supplement use were collected and those taking anti-inflammatory or lipid-lowering medications were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2010-06-01 (Actual); Primary Completion 2011-05-31 (Actual); Study Completion 2011-05-31 (Actual)

PRIMARY OUTCOMES:
serum uric acid | 4 weeks
  Hyperuricemia contributes to gout, a frequently occurring, complex rheumatologic form of inflammatory arthritis. The primary outcome measure of this study was serum uric acid and its reduction by TCJ consumption.

SECONDARY OUTCOMES:
High sensitivity C-reactive protein (hsCRP) | 4 weeks
  Elevated levels of hsCRP indicate inflammation. Serum levels of hsCRP as a secondary outcome measure were measured and the effect of TCJ in potentially lowering.
Serum triglycerides | 4 weeks
  Increased serum triglycerides contribute to CVD and MetS. Serum TG was measured as a secondary outcome measure and the effect of TCJ in lowering levels.

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Martin, PhD, MTox, Principal Investigator — Principal Investigator, School of Health Studies

IPD SHARING:
Plan to Share IPD: Yes
Coded data will be available upon reasonable request as instructed by journal editors. Emails may be directed to the Principal Investigator.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Martin KR, Coles KM. Consumption of 100% Tart Cherry Juice Reduces Serum Urate in Overweight and Obese Adults. Curr Dev Nutr. 2019 Feb 25;3(5):nzz011. doi: 10.1093/cdn/nzz011. eCollection 2019 May. PMID 31037275